CLINICAL TRIAL: NCT00832494
Title: An Open Label, Randomized, Phase I/II Study of DMXAA in Combination With Carboplatin and Paclitaxel in Patients With Locally Advanced and Metastatic Non-Small Cell Lung Cancer
Brief Title: Phase II Study of DMXAA (ASA404) in Combination With Chemotherapy in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Antisoma Research (Industry)
Responsible Party: Gary Acton, Chief Medical Officer, Antisoma Research Limited
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AS1404-201
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vadimezan; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: DMXAA in combination with carboplatin and paclitaxel — Administered every 21 days
  Other Names: DMXAA is now known as ASA404

SUMMARY:
This study was designed to test the addition of DMXAA (now known as ASA404) to carboplatin and paclitaxel in patients with NSCLC.

DETAILED DESCRIPTION:
The study was designed to determine the safety, tolerability and efficacy of DMXAA in combination with carboplatin and paclitaxel in patients with locally advanced and metastatic (Stage IIIb and IV) non-small cell lung cancer. The phase Ib part of the study evaluated dose levels of DMXAA at 600 mg/m2, 1200 mg/m2 and 1800 mg/m2. In the phase II part of the study, patients were randomized to receive carboplatin and paclitaxel alone or in combination with ASA404 1200 mg/m2. An additional single-arm study was undertaken to evaluate further patients at the 1800 mg/m2 dose level.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Histologically confirmed non-small cell lung carcinoma designated as adenocarcinoma (including bronchoalveolar), squamous cell carcinoma or undifferentiated, mixed (adenocarcinoma and squamous) or large cell carcinoma.
2. Locally advanced Stage IIIb disease, not curable with surgery or radiotherapy, or Stage IV disease.
3. Aged ≥ 18 years of age.
4. Karnofsky performance status of ≥ 70%.
5. Life expectancy of ≥ 3 months.
6. Hematological and biochemical indices at screening comprising:

   * An absolute neutrophil count of ≥ 2.0 x 109/L.
   * A platelet count of ≥ 100 x 109/L.
   * A hemoglobin level of ≥ 10 g/dL.
   * Adequate hepatic and renal function as defined by serum bilirubin ≤ 25 µmol/L; alkaline phosphatase, alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 times the upper limit of normal if no demonstrable liver metastasis or ≤ 5 times the upper limit of normal in the presence of liver metastasis; serum creatinine ≤ 120 µmol/L.
7. At least one unidimensionally measurable lesion according to the Response Evaluation Criteria in Solid Tumours (RECIST).
8. Providing written informed consent and be able to comply with study assessments and follow-up.

EXCLUSION CRITERIA:

1. Patients who had undergone major surgery, chemotherapy or radiation therapy (except palliative) within the previous 4 weeks.
2. A known history of hypersensitivity to carboplatin, paclitaxel or any of their excipients.
3. Previous exposure to DMXAA or other vascular targeting agents.
4. Small cell lung cancer or mixed histology.
5. Having received blood transfusions or growth factors to aid haematological recovery within 2 weeks of the scheduled baseline visit.
6. Active serious infection within 2 weeks of screening.
7. Clinically significant cardiac arrhythmias and known QTc prolongation.
8. Evidence of severe or uncontrolled systemic disease that might interfere with study participation.
9. A history of alcoholism, drug addiction or any psychiatric condition that would impair the patient's ability to comply with study procedures.
10. Pregnant or lactating women and women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test.
11. Patients should not have received within the two weeks prior to starting the study or be expected to need during the study period medications known to affect the QT interval or systemic serotonin levels.
12. Concurrent or previous malignancy of a different tumor type within 5 years of starting the study, except for adequately treated non-melanoma skin cancer or cervical intraepithelial neoplasia.
13. Clinical or radiological evidence of central nervous system metastases.
14. Evidence of any other clinically significant disorder or laboratory finding that might compromise patient safety.
15. Participation in any investigational drug study in which the study drug did not subsequently obtain a product license.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2004-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of combination
Tumor response rate
Time to tumor progression
Duration of response and stable disease; median and one-year survival

CONTACTS AND LOCATIONS:
Overall Officials: Mark McKeage, Principal Investigator — Auckland Medical School, Auckland, New Zealand

REFERENCES:
- [Derived] McKeage MJ, Jameson MB; AS1404-201 Study Group Investigators. Comparative outcomes of squamous and non-squamous non-small cell lung cancer (NSCLC) patients in phase II studies of ASA404 (DMXAA) - retrospective analysis of pooled data. J Thorac Dis. 2010 Dec;2(4):199-204. doi: 10.3978/j.issn.2072-1439.2010.02.04.1. PMID 22263047